CLINICAL TRIAL: NCT05265312
Title: Implementation and Evaluation of a Diabetes Prevention Clinical Pathway in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00313490; K23DK118205 (NIH)
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: PreDiabetes; Prediabetic State
Keywords: Diabetes prevention; Primary care; Clinical pathway; Pragmatic intervention
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention clinic (Active Comparator): Patients with prediabetes seen for routine care at intervention clinic
  Interventions: Other: START diabetes prevention clinical pathway
- Control clinic (No Intervention): Patients with prediabetes seen for routine care at control clinic

INTERVENTIONS:
Other: START diabetes prevention clinical pathway — The diabetes prevention clinical pathway will focus on the following steps:
  1. Screen/test - testing of eligible patients for prediabetes/diabetes
  2. Education - PCPs will be encouraged to take an online learning module and in-person group training on prediabetes management and patients with prediabetes will receive a handout about prediabetes prior to their upcoming PCP visit
  3. Action - PCPs will use a shared decision-making guide and treatment algorithm to discuss options with patients at their visit
  4. Referral - patients may be referred to DPPs and/or medical nutrition therapy (MNT)
  5. Treat - patients will be scheduled for a follow-up visit within 3-9 months with their PCP or care team to continue addressing prediabetes.
  Arms: Intervention clinic

SUMMARY:
Prediabetes is a significant public health problem affecting 88 million U.S. adults. Evidence suggest that the vast majority of people with prediabetes are unaware of having this condition and many are not receiving appropriate care for prediabetes, including referral to evidence-based programs like the Diabetes Prevention Programs (DPP). In the investigator's retrospective cohort study of patients with prediabetes from Johns Hopkins Health Systems, the investigators found that the rates of prediabetes clinical care activities are low. In the investigators' qualitative studies, the investigators found that primary care physician (PCP) barriers include low knowledge about Diabetes Prevention Programs and misperceptions of insurance coverage of these programs and inadequate clinical staff to address prediabetes. Common patient barriers to taking action to prevent diabetes include lack of motivation, time and resources.

Based on prior research, comprehensive strategies are urgently needed to improve prediabetes care. Using these findings, the investigators have designed and plan to implement a diabetes prevention clinical pathway which seeks to address some of these common clinician and patient barriers. The investigators hypothesize that the clinical pathway will result in increased clinician screening and intervention and improve patient engagement in diabetes prevention. The investigators will compare results from the intervention clinic compared to a control clinic. If successful, the investigators plan to implement and test the effectiveness of this clinical pathway across the entire health system.

ELIGIBILITY:
Inclusion Criteria:

* Prediabetes based on prediabetes registry
* Age ≥ 18 years
* PCP visit during intervention period
* Patient of Johns Hopkins Green Spring Station (GSS) General Internal Medicine or Johns Hopkins Community Physicians (JHCP) Internal Medicine clinic.

Exclusion Criteria:

* Visit with clinician who's not their Primary Care Physician (PCP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1910 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Tseng, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins General Internal Medicine clinic at Green Spring Station, Lutherville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Clinic: Patients with prediabetes seen for routine care at intervention clinic
  START diabetes prevention clinical pathway: The diabetes prevention clinical pathway will focus on the following steps:
  1. Screen/test - testing of eligible patients for prediabetes/diabetes
  2. Education - Primary Care Physicians (PCPs) will be encouraged to take an online learning module and in-person group training on prediabetes management and patients with prediabetes will receive a handout about prediabetes prior to their upcoming PCP visit
  3. Action - PCPs will use a shared decision-making guide and treatment algorithm to discuss options with patients at their visit
  4. Referral - patients may be referred to Diabetes Prevention Program (DPP) and/or medical nutrition therapy (MNT)
  5. Treat - patients will be scheduled for a follow-up visit within 3-9 months with their PCP or care team to continue addressing prediabetes.
Period: Overall Study
Arm/Group | Intervention Clinic | Control Clinic
Started | 873 | 1037
Completed | 873 | 1037
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Clinic: START diabetes prevention clinical pathway
- Control Clinic: Routine usual care
- Total: Total of all reporting groups
Arm/Group | Intervention Clinic | Control Clinic | Total
Number analyzed (Participants) | 873 | 1037 | 1910
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (13.6) | 60.7 (14.6) | 61.6 (14.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 545 | 617 | 1162
  Male | 327 | 420 | 747
  Non-binary | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 26 | 45
  Not Hispanic or Latino | 825 | 977 | 1802
  Unknown or Not Reported | 29 | 34 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 62 | 93 | 155
  Black/African American | 220 | 280 | 500
  Other | 33 | 49 | 82
  Unknown/Declined to Answer | 14 | 11 | 25
  White | 544 | 604 | 1148

OUTCOME MEASURES:

1. Primary Outcome: Number of PCP Visits Where Ppt Was Referred to Diabetes Prevention Program Within 30 Days of Visit
Description: Number of PCP visits where ppt referred to Diabetes Prevention Program during intervention period
Time Frame: 12 months
Measure: Number; unit: pcp visits
Units Other Than Participants: pcp visits
Arm/Group | Intervention Clinic | Control Clinic
Number analyzed (Participants) | 873 | 1037
Number analyzed (pcp visits) | 1754 | 2328
pcp visits | 47 | 10

2. Primary Outcome: Number of PCP Visits Where Ppt Was Prescribed Metformin Within 30 Days
Time Frame: 12 months
Measure: Number; unit: pcp visits
Units Other Than Participants: pcp visits
Arm/Group | Intervention Clinic | Control Clinic
Number analyzed (Participants) | 873 | 1037
Number analyzed (pcp visits) | 1754 | 2328
pcp visits | 58 | 39

3. Primary Outcome: Number of PCP Visits Where Ppt Was Referred to Medical Nutrition Therapy Within 30 Days
Time Frame: 12 months
Measure: Number; unit: pcp visits
Units Other Than Participants: pcp visits
Arm/Group | Intervention Clinic | Control Clinic
Number analyzed (Participants) | 873 | 1037
Number analyzed (pcp visits) | 1754 | 2328
pcp visits | 3 | 37

4. Secondary Outcome: Number of Participants Who Complete Glycemic Lab Testing Out of Those With an Order During Intervention Period
Description: Fasting glucose or Hemoglobin A1c
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Clinic | Control Clinic
Number analyzed (Participants) | 873 | 1037
Participants | 800 | 906

5. Secondary Outcome: Achieve 5% or Greater Reduction in Weight Compared to Baseline
Description: Proportion achieving 5% or greater weight reduction
Time Frame: Baseline and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Clinic | Control Clinic
Number analyzed (Participants) | 873 | 1037
Participants | 49 | 43

ADVERSE EVENTS:
Description: Adverse event data not collected
Arm/Group | Intervention Clinic | Control Clinic
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT05265312/Prot_SAP_000.pdf